CLINICAL TRIAL: NCT00939679
Title: ERGEM: Effect of Roux-en-Y Gastric Bypass Surgery on Energy Metabolism.
Brief Title: Effect of Gastric Bypass Surgery on Energy Metabolism
Acronym: ERGEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Cambridge Weight Plan Limited (Industry)
Responsible Party: Principal Investigator, AAstrup, Head of Department, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B263
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Obesity
Keywords: obesity; bariatric surgery; energy expenditure; incretins; appetite regulation; body composition; GLP-1
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Earlier gastric bypass surgery (7 weeks) (Experimental): These patients will undergo gastric bypass surgery 7 weeks after starting a low calorie diet, and will continue the low calorie diet for 3 weeks following surgery.
  Interventions: Procedure: Roux-en-Y gastric bypass surgery; Dietary Supplement: low calorie diet (1,000 kcal/day)
- Later gastric bypass surgery (10 weeks) (Active Comparator): These patients will undergo gastric bypass surgery 10 weeks after starting a low calorie diet.
  Interventions: Procedure: Roux-en-Y gastric bypass surgery; Dietary Supplement: low calorie diet (1,000 kcal/day)

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass surgery — Briefly, RYGB is characterized first by creation of a small stomach pouch. The small intestine is then divided approximately 75 cm distal to the ligament of Treitz, creating a proximal intestinal limb that transports the secretions from the stomach remnant, liver, and pancreas, and a 'Roux' limb, that is attached to the new stomach pouch to drain consumed food. The distal end of the proximal limb is then reattached approximately 100 cm distal to the new stomach drainage site, creating a common channel where digestive enzymes mix with ingested food.
Dietary Supplement: low calorie diet (1,000 kcal/day) — Patients will consume a daily diet composed of:
  * 4 powder diet portions (Cambridge Diets, UK)
  * plain yogurt (100-125g)
  * skim milk (1L)
  * a limited variety of vegetables
  The diet will be consumed by both groups for a 10 week period.
  Other Names: Cambridge Weight Plan, Northants, UK.

SUMMARY:
The purpose of this study is to investigate the short term and long term effects of Roux-en-Y gastric bypass (RYGB) surgery on energy expenditure, gastrointestinal and appetite regulating hormone levels, and appetite sensation. We hypothesize that following RYGB surgery, metabolism will be elevated in comparison to patients who have not yet had RYGB but who are losing weight simultaneously using a low calorie diet. We further hypothesize that this higher metabolism will be associated with alterations in fasting and postmeal levels of gastrointestinal and appetite regulating hormones. Long term (1.5 years after RYGB), we hypothesize that differences in metabolism, body composition, and hormone levels will distinguish between patients who have maintained their weight loss after RYGB vs those who have regained weight.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* BMI ≥40, or ≥35 with concomitant obstructive sleep apnea, or hypertension
* scheduled for RYGB surgery at Hvidovre Hospital, Copenhagen, Denmark
* Must have lost between 1-4% body weight after 3 months of dietary counselling

Exclusion Criteria:

* Deemed ineligible for RYGB surgery by patient's own physician(s)
* Diabetes Mellitus
* Non Caucasian
* Weight >160kg (due to DEXA scanner limitations), or morphologically unable to accommodate in DEXA scanner (>40cm in maximum supine anterior-posterior dimension, or >60cm in maximum supine body width)
* Hemoglobin <7.0 mmol/L
* Psychiatric illness under the care of a psychiatrist
* Eating disorder such as bulimia
* Patients on special diets (eg vegetarian, Atkins)
* Any history of thyroid dysfunction, or use of thyroid medication (with the exception of transient thyroiditis)
* Hypothalamic or genetic etiology of obesity
* A current diagnosis of cancer
* Any surgery other than RYGB planned in the ensuing 3 months
* Substance abuse or smoking
* Use of prescription medications or over-the-counter drugs affecting metabolism
* Excessive intake of alcohol (>7 drinks/week)
* Excessive intake of caffeine (>300 mg/day)
* Presence of any contraindication to use of a low calorie powder diet, including:

  * Past history of ventricular arrhythmias (even if treated)
  * Renal dysfunction (creatinine clearance <60 mL/min)
  * Liver enzymes (ALT or AST) >3x upper limit of normal
  * Milk protein allergy, or lactose intolerance
  * Porphyria or phenylketonuria
  * History of gout
  * Breastfeeding
  * Concomitant use of monoamine oxidase inhibitors or non potassium sparing diuretics
  * Inability or unwillingness to comply with a low calorie diet protocol
  * Patients who find the powder diet products to be unpalatable
* Do not enjoy yogurt, carrots, or milk (as these are essential elements of the low calorie diet)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in 24 hour energy expenditure | 7 weeks, 10 weeks (short term); 1.5 years (long term)

SECONDARY OUTCOMES:
change in fasting bile acids and lipid profile | 7 weeks, 10 weeks (short term); 1.5 years (long term)
changes in fasting levels of leptin, adiponectin, and visfatin | 7 weeks, 10 weeks (short term); 1.5 years (long term)
change in body composition | 7 weeks, 10 weeks (short term); 1.5 years (long term)
Change in appetite sensation | 7 weeks, 10 weeks (short term); 1.5 years (long term)
change in fasting and postprandial levels of GLP-1, PYY, oxyntomodulin, glucose, insulin, C peptide, GIP, ghrelin, cholecystokinin | 7 weeks, 10 weeks (short term); 1.5 years (long term)

CONTACTS AND LOCATIONS:
Overall Officials: Julie B Schmidt, MSc, Principal Investigator — University of Copenhagen
Locations (2):
- Denmark (2):
  - Department of Human Nutrition, Faculty of Life Sciences, University of Copenhagen, Copenhagen
  - Hvidovre Hospital, Copenhagen